CLINICAL TRIAL: NCT04947618
Title: Evaluation of the Efficacy of Management of Patients With Lymphomas Diagnosed at Nimes University Hospital Over 20 Years (1999-2018) Under Real-life Circumstances
Brief Title: Efficacy of Patient Management for Lymphoma Diagnosed at Nimes University Hospital From 1999 to 2018. DVR-Lym-Nim
Acronym: DVR-Lym-Nim
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2019-01/EJ-01
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma, Malignant
Keywords: -Lymphoma; Mantle-Cell; Follicular; Hodgkin; T-cell; Primitive Cerebral; Marginal Zone; Waldenström's macroglobulinemia
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Lymphoma protocol was applied. Biopsies of lymphomas used for anatomopathological analysis, frozen and used for cytogenetic analysis if possible.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observation of a cohort of 400 patients with different types of lymphomas.

DETAILED DESCRIPTION:
A database on 400 patients diagnosed with lymphomas was built up over 20 years at Nîmes University Hospital. Biopsies were made on these tumours and all the samples were frozen.

Considering the heterogeneous nature of lymphomas, randomized clinical trials based on very precise criteria for the inclusion or non-inclusion of patients are the gold standard for studying the various sub-types of lymphomas by concentrating on homogeneous populations for which a limited number of parameters are analyzed simultaneously. However, due to the complexity of their medical situation, many patients may be excluded form these trials, thus making it difficult to obtain reliable results.

The analysis of a non-selected cohort has two main advantages: (1) to better understand the diversity of patients with lymphomas for which the recommendations are constantly evolving and (2) to analyze how, exactly, these are managed by integrating points which are currently poorly evaluated such as comorbidities and accessibility to treatment.

The aim of the study is to describe how these patients are managed and to demonstrate that not all patients are able to benefit from the official management recommendations applicable to their pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 15 years and 3 months, diagnosed with lymphoma at Nîmes University Hospital as from 1999 onwards and for whom diagnostic tumor material is available.

Exclusion Criteria:

* Patients aged 18 or over who have expressed their desire not to take part in the study.
* Patients under the age of 18 whose legal representatives have expressed their desire for the child not to take part in the study.
* Patients under legal guardianship.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population consists of patients with lymphomas (Malignant Non-Hodgkinien and Hodgkin Lymphomas) diagnosed at Nîmes University Hospital from 1999 onwards and for whom the frozen biological samples are available. Since 2005, all patients have been registered in the Tumototek software program. Those diagnosed before this date can be found in the hospital's anatomopathological laboratory registers.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate among patients with Hodgkin Lymphomas | 2 years after inclusion
  The number of months during which the patient has survived since inclusion will be noted. If the patient has died, the date of death recorded in the hospital file or from the INSERM CépiDC register will be noted.
Overall survival rate among patients with Mantle-cell Lymphomas | 2 years after inclusion
  The number of months during which the patient has survived since inclusion will be noted.If the patient has died, the date of death recorded in the hospital file or from the INSERM CépiDC register will be noted.
Overall survival rate among patients with Primitive Cerebral Lymphomas | 2 years after inclusion
  The number of months during which the patient has survived since inclusion will be noted. If the patient has died, the date of death recorded in the hospital file or from the INSERM CépiDC register will be noted.
Overall survival rate among patients with Follicular Lymphomas | 2 years after inclusion
  The number of months during which the patient has survived since inclusion will be noted. If the patient has died, the date of death recorded in the hospital file or from the INSERM CépiDC register will be noted.
Overall survival rate among patients with Marginal Zone Lymphomas | 2 years after inclusion
  The number of months during which the patient has survived since inclusion will be noted. If the patient has died, the date of death recorded in the hospital file or from the INSERM CépiDC register will be noted.
Overall survival rate among patients with Waldenström's Disease | 2 years after inclusion
  If the patient has died, the date of death recorded in the hospital file or from the INSERM CépiDC register will be noted.

SECONDARY OUTCOMES:
Differences between management of patients with Hodgkin Lymphomas actually observed and data described in the literature. | 2 years after inclusion
  The actual management of these patients will be compared with the data in the literature and any differences will be noted.
Differences between management of patients with Mantle-cell Lymphomas and data described in the literature. | 2 years after inclusion
  The actual management of these patients will be compared with the data in the literature and any differences will be noted.
Differences between management of patients with Primitive Cerebral Lymphomas and data described in the literature. | 2 years after inclusion
  The actual management of these patients will be compared with the data in the literature and any differences will be noted.
Differences between management of patients with Follicular Lymphomas and data described in the literature. | 2 years after inclusion
  The actual management of these patients will be compared with the data in the literature and any differences will be noted.
Differences between management of patients with Marginal Zone Lymphomas and data described in the literature. | 2 years after inclusion
  The actual management of these patients will be compared with the data in the literature and any differences will be noted.
Differences between management of patients with Waldenström's Disease and data described in the literature. | 2 years after inclusion
  The actual management of these patients will be compared with the data in the literature and any differences will be noted.
Reasons for differences between management of patients with Hodgkin Lymphomas actually observed and data described in the literature. | 2 years after inclusion
  The reasons for any differences noted will be analyzed
Reasons for differences between management of patients with Mantle-cell Lymphomas actually observed and data described in the literature. | 2 years after inclusion
  The reasons for any differences noted will be analyzed
Reasons for differences between management of patients with Primitive Cerebral Lymphomas actually observed and data described in the literature. | 2 years after inclusion
  The reasons for any differences noted will be analyzed
Reasons for differences between management of patients with Follicular Lymphomas actually observed and data described in the literature. | 2 years after inclusion
  The reasons for any differences noted will be analyzed
Reasons for differences between management of patients with Marginal Zone Lymphomas actually observed and data described in the literature. | 2 years after inclusion
  The reasons for any differences noted will be analyzed
Reasons for differences between management of patients with Waldenström's Disease actually observed and data described in the literature. | 2 years after inclusion
  The reasons for any differences noted will be analyzed
Analysis of the efficacy of treatment of patients with Hodgkin Lymphomas. | 2 years after inclusion
  The following criteria for efficacy will be noted: overall survival, relapse, survival without relapse and refractory lymphomas. The histological type, treatment given and comorbidities noted will be included in the analysis.
Analysis of the efficacy of treatment of patients with Mantle-cell Lymphomas | 2 years after inclusion
  The following criteria for efficacy will be noted: overall survival, relapse, survival without relapse and refractory lymphomas. The histological type, treatment given and comorbidities noted will be included in the analysis.
Analysis of the efficacy of treatment of patients with Primitive Cerebral Lymphomas | 2 years after inclusion
  The following criteria for efficacy will be noted: overall survival, relapse, survival without relapse and refractory lymphomas. The histological type, treatment given and comorbidities noted will be included in the analysis.
Analysis of the efficacy of treatment of patients with Follicular Lymphomas | 2 years after inclusion
  The following criteria for efficacy will be noted: overall survival, relapse, survival without relapse and refractory lymphomas. The histological type, treatment given and comorbidities noted will be included in the analysis.
Analysis of the efficacy of treatment of patients with Marginal Zone Lymphomas | 2 years after inclusion
  The following criteria for efficacy will be noted: overall survival, relapse, survival without relapse and refractory lymphomas. The histological type, treatment given and comorbidities noted will be included in the analysis.
Analysis of the efficacy of treatment of patients with Waldenström's Disease | 2 years after inclusion
  The following criteria for efficacy will be noted: overall survival, relapse, survival without relapse and refractory lymphomas. The histological type, treatment given and comorbidities noted will be included in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Chair — CHU de Nîmes (Nîmes University Hospital)
Locations (1):
- CHU Nimes, Nîmes, France